CLINICAL TRIAL: NCT02446938
Title: A Simple Method for Confirming the Optimal Position of Esophageal Balloon in Patients With Mechanical Ventilation
Brief Title: Position of Esophageal Balloon in Patients With Mechanical Ventilation
Status: Completed | Type: Observational
Sponsor: Capital Medical University (Other)
Collaborators: Beijing Municipal Administration of Hospitals (Other Government)
Responsible Party: Principal Investigator, Jian-Xin Zhou, Professor, Capital Medical University
Other Study IDs: KY-2015-CCM-002
Record Dates: First submitted 2015-05-14; First posted 2015-05-18 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-06

CONDITIONS: Mechanical Ventilation
Keywords: mechanical ventilation; esophageal pressure; catheter position; validation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Esophagus balloon catheter insertion. — Esophagus balloon catheter will be inserted and the position of the balloon will be confirmed by a air injection test.A bolus of 30 ml of air was injected to the gastric lumen of the catheter just next to the distal edge of the balloon, during the onset of end-expiratory phase. The presence of a positive disturbing wave (PDW) in esophageal pressure waveform to this air injection will be the indicator of the right balloon position.

SUMMARY:
Transpulmonary pressure is frequently monitored in patients with mechanical ventilation. Right position of the catheter balloon is the key factor in accurate measurement. A simple method for confirming the balloon position will be validate in this study.

DETAILED DESCRIPTION:
Transpulmonary pressure, which is the pressure at the airway opening minus pleural pressure, is frequently monitored in patients with mechanical ventilation. Because pleural pressure is difficult to measure in most clinical situations, esophageal pressure (Pes) is used as a surrogate. Catheter with air balloon is the most commonly used method to measure the Pes. Right position of the balloon is the key factor in accurate measurement of Pes, and the lower third part of esophagus is recommended as the target position of the balloon. The catheter is usually inserted into the stomach first, and then slowly withdrawn into the esophagus after inflation of the balloon. A negative pressure deflection replacing the positive pressure deflection during inspiration generally indicates the balloon's entering into the esophagus. This confirmation method depends on the normal function of diaphragm. However, it may not always be possible to obtain the standard pressure deflections in patients with mechanical ventilation, especially in those with diaphragmatic paralysis.

In present study, the investigators developed a simple method to confirm the balloon position by using a modified SmartcathG esophageal balloon catheter. The objective was to evaluate the validity of this method and to investigate the relationship between the cardiac artifacts of the Pes tracings and the position of the balloon.

ELIGIBILITY:
Inclusion Criteria:

* adult patients receiving invasive mechanical ventilation

Exclusion Criteria:

* age under 18 years old
* esophageal varices
* evidence of active air leak from the lung, including bronchopleural fistula, pneumothorax, pneumomediastinum, or existing chest tube
* history of chronic obstructive pulmonary disease
* history of lung surgery
* pregnancy
* severe coagulopathy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with mechanical ventilation.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-05; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
The agreement of balloon position confirmed by air injection method and confirmed by the bed-side X-ray. | 15 min after the balloon position

CONTACTS AND LOCATIONS:
Locations (1):
- ICU, Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Chen H, Xu M, Yang Y, He X, Zhou J. [Application of injection test in confirming the ideal position of esophageal balloon catheter]. Zhonghua Wei Zhong Bing Ji Jiu Yi Xue. 2017 Sep;29(9):783-788. doi: 10.3760/cma.j.issn.2095-4352.2017.09.004. Chinese. PMID 28936952